CLINICAL TRIAL: NCT00775944
Title: Trial Comparing Different Methods of Support With Stopping Smoking Offered Through The National Health Service (NHS) Smoking Helpline
Brief Title: Trial Comparing Different Methods of Support With Stopping Smoking (PORTSSS/Stop Together Trial)
Acronym: PORTSSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Department of Health, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 08118
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-09

CONDITIONS: Tobacco Smoking
Keywords: Tobacco; Cigarette; Smoking; Counselling; Nicotine Replacement Therapy; Telephone; Quitline; Helpline
MeSH Terms: conditions — Tobacco Smoking; Smoking | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard support (Active Comparator): Standard 'Together Programme' telephone support for smoking cessation & advice to obtain nicotine addiction treatment
  Interventions: Behavioral: Reactive (standard) telephone support
- Proactive telephone support (Active Comparator): Proactive support & advice to obtain nicotine addiction treatment
  Interventions: Behavioral: Proactive telephone support
- Standard support & offer NRT (Active Comparator): Reactive telephone support (i.e. Together Programme) and offer of voucher for cost free Nicotine Replacement Therapy
  Interventions: Behavioral: Reactive (standard) telephone support; Drug: Offer of voucher for cost-free Nicotine Replacement Therapy
- Proactive support & offer NRT (Active Comparator): Proactive telephone support and offer of voucher for cost free NRT
  Interventions: Behavioral: Proactive telephone support; Drug: Offer of voucher for cost-free Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Proactive telephone support — Pro-active telephone counselling allows for repeated, sequenced calls to be made by quitline counsellors to smokers and for counselling to be provided during accepted calls.
  Other Names: Telephone; Counselling
  Arms: Proactive support & offer NRT; Proactive telephone support
Behavioral: Reactive (standard) telephone support — Reactive counselling usually involves the provision of evidence-based information to support quit attempts without any or with only very brief counselling to accompany it.
  Other Names: Together Programme
  Arms: Standard support; Standard support & offer NRT
Drug: Offer of voucher for cost-free Nicotine Replacement Therapy — Offer of voucher for cost-free Nicotine Replacement Therapy over the telephone
  Other Names: NRT
  Arms: Proactive support & offer NRT; Standard support & offer NRT

SUMMARY:
This study shall determine whether or not proactive telephone support for smoking cessation delivered to quitline callers is more effective than standard 'reactive' provision and whether or not the offer of a voucher for a cost free supply of nicotine replacement therapy (NRT) has any additional impact on smoking cessation rates achieved by behavioural interventions.

DETAILED DESCRIPTION:
There is evidence from other studies that telephone helplines are effective in helping individuals to stop smoking. This study will investigate whether or not two interventions that have been proven effective in other contexts are effective when offered via telephone helplines. The two interventions which will be tested are (1) additional proactive counselling via telephone(several calls from a trained smoking cessation advisor over a certain period) and (2) the offer of Nicotine Replacement Therapy.

This trial will determine whether or not: (1)additional (proactive) telephone support for smoking cessation delivered to users of the National Health Service (NHS)Smoking Helpline, is more effective than standard support given by the helpline, and (2) whether the offer of free Nicotine Replacement Therapy influences rates of stopping smoking in individuals receiving either standard (reactive) or proactive telephone support.

Current smokers over 16 years of age will be recruited by helpline staff with the appropriate consent. Participants will then be randomised into one of four groups:

(i) usual care delivered by the helpline (called the Together Programme) (ii) usual care plus a programme of proactive telephone counselling (iii) usual care AND the offer of Nicotine Replacement Therapy (NRT) (iv) usual helpline support, proactive telephone counselling AND the offer of NRT.

The researchers will not be aware of which group participants have been allocated. The results will determine if the use of proactive telephone counselling is effective in helping individuals to stop smoking. It shall also find out if the offer of NRT medication via a telephone helpline assists individuals in their efforts to stop smoking.

ELIGIBILITY:
Inclusion Criteria:

* Participants are over 16 and will need to agree to i) receive counselling ii) to set a quit within two weeks and iii) consent to follow up processes.

Exclusion Criteria:

* Telephonists will not enrol potential participants who are not capable of giving informed consent or who have not got access to a phone contact number to which calls can be made by Essentia staff.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2591 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Coleman, MB ChB, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Background] Silagy C, Mant D, Fowler G, Lancaster T. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2000;(3):CD000146. doi: 10.1002/14651858.CD000146. PMID 10908462
- [Background] Tobacco Advisory Group of the Royal College of Physicians. Going smoke-free: The case for clean air in the home, at work and in public places. London: Royal College of Physicians of London, 2005.
- [Background] Tobacco Advisory Group of the Royal College of Physicians. Nicotine addiction in Britain. London: Royal College of Physicians of London, 2000.
- [Background] Ashenden R, Silagy C, Weller D. A systematic review of the effectiveness of promoting lifestyle change in general practice. Fam Pract. 1997 Apr;14(2):160-76. doi: 10.1093/fampra/14.2.160. PMID 9137956
- [Background] Pierce JP, White MM, Gilpin EA. Adolescent smoking decline during California's tobacco control programme. Tob Control. 2005 Jun;14(3):207-12. doi: 10.1136/tc.2004.010116. PMID 15923472
- [Background] Hughes JR, Stead LF, Lancaster T. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2000;(4):CD000031. doi: 10.1002/14651858.CD000031. PMID 11034670
- [Background] Tonstad S, Tonnesen P, Hajek P, Williams KE, Billing CB, Reeves KR; Varenicline Phase 3 Study Group. Effect of maintenance therapy with varenicline on smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):64-71. doi: 10.1001/jama.296.1.64. PMID 16820548
- [Background] Ferguson J, Bauld L, Chesterman J, Judge K. The English smoking treatment services: one-year outcomes. Addiction. 2005 Apr;100 Suppl 2:59-69. doi: 10.1111/j.1360-0443.2005.01028.x. PMID 15755262
- [Background] Stead LF, Lancaster T. Group behaviour therapy programmes for smoking cessation. Cochrane Database Syst Rev. 2000;(2):CD001007. doi: 10.1002/14651858.CD001007. PMID 10796582
- [Background] Lancaster T, Stead LF. Individual behavioural counselling for smoking cessation (Cochrane Review). The Cochrane Library, Issue 4, Chichester, UK: John Wiley & Sons, Ltd, 2003.
- [Background] Coleman T, Lewis S, Hubbard R, Smith C. Impact of contractual financial incentives on the ascertainment and management of smoking in primary care. Addiction. 2007 May;102(5):803-8. doi: 10.1111/j.1360-0443.2007.01766.x. PMID 17506157
- [Background] Britton J, Lewis S. Trends in the uptake and delivery of smoking cessation services to smokers in Great Britain. J Epidemiol Community Health. 2004 Jul;58(7):569-70. doi: 10.1136/jech.2003.015271. No abstract available. PMID 15194717
- [Background] Stead LF, Lancaster T, Perera R. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2003;(1):CD002850. doi: 10.1002/14651858.CD002850. PMID 12535442
- [Background] Platt S, Tannahill A, Watson J, Fraser E. Effectiveness of antismoking telephone helpline: follow up survey. BMJ. 1997 May 10;314(7091):1371-5. doi: 10.1136/bmj.314.7091.1371. PMID 9161308
- [Background] An LC, Schillo BA, Kavanaugh AM, Lachter RB, Luxenberg MG, Wendling AH, Joseph AM. Increased reach and effectiveness of a statewide tobacco quitline after the addition of access to free nicotine replacement therapy. Tob Control. 2006 Aug;15(4):286-93. doi: 10.1136/tc.2005.014555. PMID 16885577
- [Background] Silagy C, Lancaster T, Stead L, Mant D, Fowler G. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2002;(4):CD000146. doi: 10.1002/14651858.CD000146. PMID 12519537
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Ferguson J, Docherty G, Bauld L, Lewis S, Lorgelly P, Boyd KA, McEwen A, Coleman T. Effect of offering different levels of support and free nicotine replacement therapy via an English national telephone quitline: randomised controlled trial. BMJ. 2012 Mar 23;344:e1696. doi: 10.1136/bmj.e1696. PMID 22446739
- [Derived] Coleman T, McEwen A, Bauld L, Ferguson J, Lorgelly P, Lewis S. Protocol for the Proactive Or Reactive Telephone Smoking CeSsation Support (PORTSSS) trial. Trials. 2009 Apr 28;10:26. doi: 10.1186/1745-6215-10-26. PMID 19400961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 2009 and January 2010. 2591 participants were randomised to one of the four treatment groups. Of these, 56 withdrew consent after being randomised and were not included in analyses.
Groups:
- Standard Support & Offer of NRT: Reactive telephone support (i.e. Together Programme) and offer of voucher for cost free Nicotine Replacement Therapy
- Proactive Support & Offer of NRT: Proactive telephone support and offer of voucher for cost free NRT
Period: Overall Study
Arm/Group | Standard Support | Standard Support & Offer of NRT | Proactive Telephone Support | Proactive Support & Offer of NRT
Started | 648 | 647 | 648 | 648
Completed | 633 (15 participants withdrew consent) | 638 (9 participants withdrew consent) | 632 (16 participants withdrew consent) | 632 (16 participants withdrew consent)
Not Completed | 15 | 9 | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT | Total
Number analyzed (Participants) | 648 | 648 | 647 | 648 | 2591
Age Continuous [Mean (Standard Deviation); unit: years] | 40.3 (14.5) | 39.7 (14.8) | 38.6 (14.8) | 39.6 (14.1) | 39.6 (14.5)
Age, Customized [Number; unit: participants]
  < 18 years | 12 | 14 | 13 | 11 | 50
  18-64 years | 569 | 562 | 564 | 575 | 2270
  >=65 years | 33 | 41 | 44 | 31 | 149
  Unknown | 34 | 31 | 26 | 31 | 122
Sex/Gender, Customized [Number; unit: participants]
  Female | 328 | 321 | 350 | 356 | 1355
  Male | 293 | 301 | 275 | 268 | 1137
  Unknown | 27 | 26 | 22 | 24 | 99
Region of Enrollment [Number; unit: participants]
  United Kingdom | 648 | 648 | 647 | 648 | 2591

OUTCOME MEASURES:

1. Primary Outcome: Self-reported, Prolonged Abstinence From Smoking Between a Quit Date and 6 Months Afterwards.
Description: Prolonged abstinence was defined as not smoking between a quit date and six months later with minor smoking lapses permitted as long as no more than 5 cigarettes in total were smoked during this period.
Time Frame: 6 months from participant's quit date
Population: All randomised cases
Measure: Number; unit: participants
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT
Number analyzed (Participants) | 648 | 648 | 647 | 648
participants | 127 | 124 | 114 | 104

2. Secondary Outcome: Self-reported Point Prevalence Abstinence From Smoking for at Least 7 Days, Ascertained at 6 Months, With Carbon Monoxide (CO) Validation.
Description: The participant had to report not smoking for at least 7 days prior to the point of outcome assessment.
Time Frame: Measured 6 months after participant's quit date
Measure: Number; unit: participants
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT
Number analyzed (Participants) | 648 | 648 | 647 | 648
participants | 62 | 57 | 42 | 39

3. Secondary Outcome: Self-reported Abstinence From Smoking for at Least Three Months, Ascertained at 6 Months
Description: Participants had to report not smoking in the three months prior to outcome ascertainment.
Time Frame: Measured at 6 months after participant's quit date
Population: All randomised cases
Measure: Number; unit: participants
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT
Number analyzed (Participants) | 648 | 648 | 647 | 648
participants | 102 | 114 | 100 | 85

4. Secondary Outcome: Self-reported Prolonged Abstinence From Smoking Between a Quit Date and 1 Month
Description: Prolonged abstinence was defined as not smoking between a quit date and one month later; minor lapses were permitted provided no more than 5 cigarettes in total had been smoked.
Time Frame: Measured at 1 month after participant's quit date
Population: All randomised cases
Measure: Number; unit: participants
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT
Number analyzed (Participants) | 648 | 648 | 647 | 648
participants | 257 | 263 | 276 | 244

5. Secondary Outcome: Self-reported Point Prevalence Abstinence From Smoking for at Least 7 Days, Ascertained at 1 Month
Description: Participants had to report not smoking for 7 or more days prior to outcome ascertainment.
Time Frame: Measured at 1 month after participant's quit date
Population: All randomised cases
Measure: Number; unit: participants
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT
Number analyzed (Participants) | 648 | 648 | 647 | 648
participants | 215 | 202 | 223 | 191

6. Secondary Outcome: Number of Unsuccessful Quit Attempts Lasting > 24 Hrs Reported at One and 6 Months
Description: As title
Time Frame: Measured 6 months after participant's quit date
Reporting Status: Not Posted

7. Secondary Outcome: Health Status at 6 Months EuroQol 5D (EQ5D)
Description: This is a generic measure of health status used in health economic analyses.
Time Frame: Measured 6 months after participant's quit date
Reporting Status: Not Posted

8. Secondary Outcome: Use of Other NHS Smoking Cessation Interventions (e.g. Uptake of NHS Stop Smoking Services, Use of Other NRT Obtained From General Practitioner (GP) Etc.)
Description: Participants' recall of the use they have made of other stop smoking interventions that are available through the National Health Service.
Time Frame: Measured 6 months after participant's quit date
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Standard Support | Proactive Telephone Support | Standard Support & Offer of NRT | Proactive Support & Offer of NRT
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No